CLINICAL TRIAL: NCT05583656
Title: INSPIRIS RESILIA Valve in Pulmonary Position - A Prospective Clinical Trial
Brief Title: INSPIRIS RESILIA Valve in Pulmonary Position
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Erhan Urganci, MD, Medical University of Vienna
Other Study IDs: 1888/2018
Record Dates: First submitted 2022-10-13; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Pulmonary Valve Disorder; Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Edwards Inspiris Resilia Valve
  Interventions: Procedure: Pulmonary valve replacement

INTERVENTIONS:
Procedure: Pulmonary valve replacement — Surgical replacement of the pulmonary valve using the Edwards Inspiris Resilia prosthesis.

SUMMARY:
In this trial we intend to evaluate the safety and effectiveness of the INSPIRIS valve prothesis in the pulmonary position in patients of five years or older, with congenital or acquired pulmonary valve disease, requiring replacement of their native or prosthetic pulmonary valve.

DETAILED DESCRIPTION:
Up to 40 subjects will be invited to participate in this trial after the indication for pulmonary valve replacement has been established. At the inclusion visit, patients will be screened according to the inclusion / exclusion criteria. After written informed consent, a detailed history will be obtained, and the study related exams will be performed.

The procedure will be performed through a median sternotomy with the help of cardiopulmonary bypass in a beating or arrested heart fashion depending on the individual surgeon's discretion. Any additional or residual defects will concomitantly be addressed. Either a native or prosthetic pulmonary valve will be replaced by an Edwards Inspiris valve (Edwards Lifesciences, Unterschleissheim, Germany). If a conduit is required, the valve will be sewn into a suitable prosthesis beforehand.

Subjects will be seen regularly after pulmonary valve implantation at hospital discharge, 6-month, 1 year and 2 years after surgery. A cardiac magnetic resonance imaging will be performed at inclusion and 2 years after surgery.

Total enrollment period for the study is estimated to be two years. The trial starts with the enrollment of the first patients and ends after the last patient enrolled has completed the two-year visit or has exited the study.

ELIGIBILITY:
Inclusion Criteria:

1. pulmonary valve disease requiring pulmonary valve replacement of their native or prosthetic valve, equal to or greater than five years of age.
2. Patients and/or patient´s legal representatives must provide written informed consent as approved and required by the respective institutional review board and agree to its provisions.
3. The patient has completed all preoperative investigations.

Exclusion Criteria:

1. Requires emergency surgery
2. Has acute myocardial infarction (MI) within 30 days prior to screening date
3. Has MRI or CT scan confirmed stroke, cerebrovascular accident (CVA) or transient ischemic attack (TIA) within six months prior to screening date
4. Has hemodynamic or respiratory instability requiring inotropic support, mechanical circulatory support, or mechanical ventilation within 30 days prior to screening date
5. Has active endocarditis/myocarditis or endocarditis/myocarditis within three months prior to screening date
6. Has renal insufficiency as determined by creatinine level ≥ 2.5 mg/dL within 60 days prior to screening visit or end-stage renal disease
7. Has documented:

   1. leukopenia (WBC < 3.5x 103/µL),
   2. acute anemia (Hgb<10.0 g/dL or 6 mmol/L), or
   3. thrombocytopenia (platelet count < 50x 103/µL) accompanied by history of bleeding diathesis or coagulopathy within 60 days prior screening date

9. Diagnosed with abnormal calcium metabolism and/or hyperparathyroidism 10. Echocardiographic evidence of an intra-cardiac mass, thrombus, or vegetation 11. RVOT aneurysm unless treated during pulmonary valve replacement surgery 12. Has prior organ transplant or is currently an organ transplant candidate 13. Was previously implanted with study trial device 14. Previously implanted with an aortic, mitral, or tricuspid bioprosthetic valve or mechanical valve 16. Has presence of non-cardiac disease limiting life expectancy to less than 12 months 17. Is currently or has recently participated (within six weeks) in another investigational drug or device trial 18. Positive urine or serum pregnancy test in female subjects of child-bearing potential and/or nursing mothers 20. Currently incarcerated or unable to give voluntary informed consent 21. Documented history of substance (drug or alcohol) abuse within the last five years prior to screening date

Ages: 5 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients with pulmonary valve disease requiring pulmonary valve replacement of their native or prosthetic valve, equal to or greater than five years of age.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-08-12 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from death and reoperation | 2 years after implantation
  The primary safety endpoint for the trial is freedom from device or procedure related death and/or reoperation at 2 years after implantation.

SECONDARY OUTCOMES:
Safety endpoints | 2 years after implantation
  all-cause mortality, structural valve deterioration, paravalvular leak, non-structural valve deterioration, transvalvular leak, trial valve-related mortality, endocarditis, valve thrombosis, explant and thromboembolism

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No